CLINICAL TRIAL: NCT04768777
Title: Behavioral Intervention for Physical Activity and Sexual Dysfunction in Multiple Sclerosis
Acronym: BIPAMS-SD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Donald Lein, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300006813
Record Dates: First submitted 2021-02-10; First posted 2021-02-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Sexual Dysfunction
Keywords: physical activity; sexual behaviour
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Sexual Dysfunction, Physiological; Motor Activity; Coitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention for Physical Activity in MS (BIPAMS) (Experimental): A behavioral intervention that involves an internet website and one-on-one video coaching calls for increasing physical activity in people with MS.
  Interventions: Behavioral: Behavioural intervention for physical activity for multiple sclerosis (BIPAMS)
- waitlist control condition (No Intervention): Participants will have 16-weeks of no intervention or interaction.

INTERVENTIONS:
Behavioral: Behavioural intervention for physical activity for multiple sclerosis (BIPAMS) — The current behavioral intervention consists of two primary components; an internet website and one-on-one video chats with a behavioral coach. The internet website involves content delivered through interactive video courses.The interactive video courses are based on elements of social cognitive theory. Each course consists of an introduction, the primary content, and a take home message.The interactive courses include embedded, supplementary options such as videos on content and worksheets related to the topic.A pedometer is provided for tracking steps, and these steps will be entered into the website so progress can be monitored. The chats support adherence to the intervention,discussion of website material,supportive accountability,and reporting of adverse events/injuries. The chats are conducted face-to-face through an online videoconferencing platform. There are a total of 12 chats over 16 weeks. Chats occur on weeks 1-8, 10-11, 13 and16.
  Arms: Behavioral Intervention for Physical Activity in MS (BIPAMS)

SUMMARY:
The prevalence of sexual dysfunction is higher among women with multiple sclerosis (MS) than women in the general population. The presence of sexual dysfunction is associated with decreased well-being and quality of life. There is limited research supporting pharmacological and other therapeutic approaches for managing sexual dysfunction in MS. Physical activity has beneﬁcial eﬀects on many of the consequences of MS, and physical activity represents a promising non-pharmacological approach for managing symptoms of sexual dysfunction in MS. The proposed research examines the eﬀect of an Internet-delivered lifestyle physical activity intervention for improving sexual dysfunction in women with MS. The research proposed, if successful, will provide evidence for the eﬃcacy of physical activity as a translatable approach for managing sexual dysfunction among women with MS.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Diagnosed of relapsing remmiting multiple sclerosis
3. Relapse free in the past 30 days
4. Initial confirmation of sexual dysfunction (based on a semi-structured interview on sexual dysfunction diagnostic criteria in DSM-5)
5. Currently in a committed relationship with a partner who does not have a sexual disorder or sexual dysfunction
6. Internet and email access
7. Willingness to complete the questionnaires, wear the pedometer, and undergo randomization
8. Insufficient physical activity [not meeting current physical activity guidelines based on a health contribution score of less than 14 units from the Godin Leisure-Time Exercise Questionnaire (GLTEQ)]
9. Ability to ambulate without assistance [self-report and Patient-Determined Disease Steps (PDDS) score between 0 and 2 (mild ambulatory disability)]
10. Age between 18 and 45 years
11. English as primary language

    -

    Exclusion Criteria:

1. Moderate or high risk for contraindications of possible injury or death when undertaking strenous or maximal exercise

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Sexual Dysfunction at 16 weeks | Baseline, week 16
  The Female Sexual Function Index (FSFI): is a common generic measure of sexual dysfunction for women. The questionnaire consists of 19 questions that cover six subscales/domains of sexual function: sexual desire, sexual arousal, lubrication, orgasm, sexual satisfaction, and pain. The items further yield an overall score. Lower sum scores reflect more pronounced sexual dysfunction.

SECONDARY OUTCOMES:
Change from baseline Sexual Dysfunction in MS at 16 weeks | Baseline, week 16
  The Multiple Sclerosis Intimacy and Sexuality Questionnaire (MSISQ-19) is the most widely used self-rating tool for sexual functions in MS (Sanders et al., 2000). The MSISQ-19 consists of 19 items focusing on the perceived influence of MS symptoms on sexual activity and satisfaction and the perceived influence of MS symptoms on the overall quality of intimate relationships. The scores classifies the type of sexual dysfunction in to primary, secondary, or tertiary sexual dysfunction.
Change from baseline Physical activity at 16 weeks | Baseline, week 16
  GLTEQ: Physical Activity Levels as measured by the Godin Leisure-Time Exercise Questionnaire. Participants will complete the Godin Leisure-Time Exercise Questionnaire (GLTEQ) as a measure of the frequency of strenuous, moderate, and mild leisure-time physical activity performed for periods of 15 minutes or more over a typical week. Summary scores are calculated by multiplying the number of strenuous, moderate, and mild bouts by 9, 5, and 3, respectively, and summing those values into an overall score that ranges from 0 to 119; higher scores are represent a greater volume of physical activity. This will be completed at baseline testing.
Change from baseline physical activity duration at 16 weeks | Baseline, week 16
  International Physical Activity Questionnaire (IPAQ). The IPAQ was developed by a working group initiated by the World Health Organization and the Centers for Disease Control and Prevention. The IPAQ asks participants about time spent in physical activity over the last seven days. Minutes of walking, sedentary-, moderate- and vigorous-intensity activities were calculated for the past week.

OTHER OUTCOMES:
Stability and changes of Fatigue over time | Baseline, week 16
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Change from Baseline Depression at 16 weeks | Baseline, week 16
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Change from Baseline Anxiety at 16 weeks | Baseline, week 16
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Change from Baseline Subjective sleep complaints at 16 weeks | Baseline, week 16
  Insomnia Severity Index (ISI). This questionnaire is a seven-item screening measure for insomnia. The items, answered on a 5-point Likert scale ranging from 0 (=not at all) to 4 (=very much), refer in part to the Diagnostic and Statistical Manual of Mental Disorders criteria for insomnia by assessing difficulty falling asleep, difficulty remaining asleep, early morning awakenings, impaired daytime performance, low satisfaction with sleep, and worry about sleep. The higher the overall score, the more the participant is assumed to suffer from insomnia.
Change from Baseline Feelings of Loneliness at 16 weeks | Baseline, week 16
  Short-form UCLA Loneliness Scale is a 3-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation.
Change from Baseline Pain severity at 16 weeks | Baseline, week 16
  Short-form of McGill Pain Questionnaire : Change of self-report measures of Pain through the Short-form of McGill Pain.
Change from Baseline Emotion Regulation at 16 weeks | Baseline, week 16
  Emotion Regulation Questionnaire(ERQ): A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Lowersscores reflects better emotion regulation.
Change from Baseline Couple Satisfaction at 16 weeks | Baseline, week 16
  Couple Satisfaction Index (CSI-4), is a seven-item questionnaire for assessing the level of couple satisfaction. The answers are given on a 7-point Likert scale (for question 1) and 6-point Likert scale (for question 2-4) with the following anchor points 0 (= extremely unhappy/not at all satisfied) to 6 or 5 (= Perfect/completely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States